CLINICAL TRIAL: NCT05258084
Title: The Effect of Sexual Minority Awareness Education Provided to Nursing Students on the Level of Knowledge and Attitudes Towards LGBT Individuals
Brief Title: The Effect of Sexual Minority Awareness Education on the Level of Knowledge and Attitude Towards LGBT Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İstanbul Yeni Yüzyıl Üniversitesi (Other)
Responsible Party: Principal Investigator, Sevcan Karataş, Lecturer, PhD Cand., Mental Health and Psychiatric Nursing, İstanbul Yeni Yüzyıl Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202107-687
Record Dates: First submitted 2022-02-11; First posted 2022-02-28 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Sexual and Gender Minorities; Attitude
Keywords: sexual minority; LGBT; attitude; education; nursing student
MeSH Terms: conditions — Coitus; Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- initiative group (Experimental): 1st and 2nd year nursing students who have not received education for sexual minorities before and continue their education at a university. Sexual minority awareness training will be applied to this group
  Interventions: Behavioral: sexual minority awareness training
- control group (No Intervention): 1st and 2nd year nursing students who have not received education for sexual minorities before and continue their education at a university. Sexual minority awareness training will not be applied to this group

INTERVENTIONS:
Behavioral: sexual minority awareness training — sexual minority awareness training is planned as 4 interviews (1 interview per week) for a total of 4 hours. Gender and sexuality-related terminologies and concepts will be discussed in the 1st meeting. Expression of sexual identity and gender transition processes will be examined in the 2nd meeting. In the 3rd meeting, the determining factors in the inadequate utilization of health services by LGBT individuals will be discussed. In the 4th meeting, what can be done to create a safe and health-friendly environment for LGBT individuals and healthcare professionals will be discussed.
  Arms: initiative group

SUMMARY:
Purpose:This research was planned to determine the effect of the sexual minority awareness training program given to nursing students on the level of knowledge and attitude towards LGBT individuals.

Design:The study was planned as an experimental study with a randomized control group, using pre-test, post-test and follow-up test. LGBT Ally Identity Measure, Attitude Towards Lesbians and Gays Scale, Attitudes Toward Transgendered Individuals Scale will be used as data collection forms.

Hypotheses:

H1: The LGBT Ally Identity Measure scores of students who receive sexual minority awareness training will increase after the training

H2: The LGBT Ally Identity Measure scores of students receiving sexual minority awareness training will increase compared to the control group.

H3: Attitude Towards Lesbians and Gays scale scores of students who receive sexual minority awareness training will increase after the training

H4: Attitude Towards Lesbians and Gays scale scores of students who receive sexual minority awareness training will increase compared to the control group.

H5: Attitudes Toward Transgendered Individuals Scale scores of students who receive sexual minority awareness training will increase after the training

H6: Attitudes Toward Transgendered Individuals Scale scores of students who receive sexual minority awareness training will increase compared to the control group.

DETAILED DESCRIPTION:
This research was planned to determine the effect of the sexual minority awareness training program given to nursing students on the level of knowledge and attitude towards LGBT individuals.

The study was planned as an experimental study with a randomized control group, using pre-test, post-test and follow-up test. LGBT Ally Identity Measure, Attitude Towards Lesbians and Gays Scale, Attitudes Toward Transgendered Individuals Scale will be used as data collection forms.

ELIGIBILITY:
Inclusion Criteria:

* Be a student of the faculty of nursing
* No barriers to accessing technology for participation in the online training program
* Absence of a communication barrier related to vision and hearing

Exclusion Criteria:

* leaving the nursing faculty for various reasons
* have received training on sexual minorities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
LGBT Ally Identity Measure | Change of LGBT Ally Identity Measure score after 2 months
  It consists of 19 items.The scale was developed to measure awareness of the subjective experiences of these individuals and the problems they experience in society, focusing on more than measuring the attitudes and knowledge levels towards individuals belonging to sexual minorities.It is in a five-point Likert type, ranging from "strongly disagree" to "strongly agree". The total score range of the scale varies between 19-95. A high score on the scale is an indication of high supportive identity characteristics.
Attitude Towards Lesbians and Gays Scale | Change of Attitude Towards Lesbians and Gays Scale score after 2 months
  It is a five-point Likert-type measurement tool consisting of 10 items.Individuals are asked to express their opinions in five levels: "I strongly disagree", "I do not agree", "I am undecided", "I agree" and "I totally agree".Six of the items against homosexuality have negative meanings and four have positive meanings. While scoring positive items, the answer "I totally agree" is scored with "5" and the answer "I strongly disagree" with "1". In scoring negative items, the answer "I strongly disagree" is scored with "5" and the answer "I totally agree" with "1". The lowest 10 points and the highest 50 points can be obtained from the scale; higher scores indicate positive attitudes towards homosexuality; low scores mean negative attitudes.
Attitudes Toward Transgendered Individuals Scale | Change of Attitudes Toward Transgendered Individuals Scale score after 2 months
  The scale is a five-point Likert type scale consisting of 20 items in total. Each item of the scale can be answered as "strongly agree", "agree", undecided", "disagree" and "strongly disagree". Items 1, 5, 8, 10, 12, 13, 14, 16 and 17 in the scale are scored inversely. As the score obtained from the scale increases, positive attitudes towards transgender individuals increase.

CONTACTS AND LOCATIONS:
Overall Officials: Sevcan Karataş, PhD Cand, Study Director — İstanbul Yeni Yüzyıl Üniversitesi
Locations (1):
- Istanbul Yeni Yuzyil University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No